CLINICAL TRIAL: NCT05874843
Title: Validation of Point-of-care Thromboelastography (TEG 6s) in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Matthew Landman, Associate Professor of Surgery, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18124
Record Dates: First submitted 2023-04-25; First posted 2023-05-25 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-05

CONDITIONS: Coagulopathy
Keywords: thromboelastography
MeSH Terms: conditions — Hemostatic Disorders | interventions — Thrombelastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pediatric Participants (Other): Pediatric surgery patients undergoing elective pediatric surgical cases under anesthesia will be invited to participate in this prospective laboratory test validation study. The results of the interventional test will not be used in clinical decision making for the participant.
  Interventions: Diagnostic Test: Thromboelastography (TEG 6S)

INTERVENTIONS:
Diagnostic Test: Thromboelastography (TEG 6S) — The TEG 6s assays are performed in a microfluidic cartridge which only requires a small amount of a patient's blood be transferred to the cartridge for analysis. The vibration frequency of the blood meniscus at which resonance occurs is used to create a clot dynamics tracing.

SUMMARY:
The goal of this observational study is to learn about the performance of the TEG6s in normal pediatric patients. The main questions it aims to answer are: What are the normal TEG 6S lab results in normal pediatric patients and how do they compare to existing published reference ranges. Participants and their guardians will be asked to submit a small amount of blood at the beginning of an elective operation for analysis in the TEG 6s machine.

DETAILED DESCRIPTION:
Trauma is the leading cause of death in children. Researchers, starting with Trunkey et al., have described three general time points of mortality after trauma - in the field, early secondary to hemorrhage and late due to infectious complications. Early mortality after trauma is specifically linked to hemorrhage. Trauma-induced coagulopathy is a multifactorial phenomenon present after trauma in both children and adults that can worsen hemorrhage and ultimately lead to increased mortality. Classical laboratory measurements of the coagulation pathway (PT, PTT, INR, fibrinogen, platelet count) have shown derangement after trauma and are correlated with mortality. However, these traditional tests of coagulation function take time to run as they are drawn and sent to a laboratory for evaluation and therefore provide a delayed snapshot of a potentially evolving coagulopathy scenario. Adult trauma centers have increasingly incorporated viscoelastic measures of the coagulation cascade to evaluate for and subsequently treat trauma-induced coagulopathy. One such test is thromboelastography (TEG) which is a whole blood assay that assesses functional clot kinetics and stability. It provides information on how various hemostatic factors, including coagulation factors, platelets, and fibrinogen, contribute to the clot. A 2016 randomized-controlled trial in adult trauma patients who met criteria for the institutions massive transfusion protocol were randomized to transfusion guided by TEG or by conventional measure of coagulopathy. The authors found increased survival in the TEG group as well as less transfusion of platelets and fresh frozen plasma.

TEG assesses the clot rate, clot strength, and clot stability, which then assists the clinician in choosing appropriate blood component therapy. The American College of Surgeons Trauma Quality Improvement Program recommends the use of thromboelastography when patients are at risk for trauma-induced coagulopathy. Visicoeslastic evaluation of the coagulation pathway has become the standard of care in adult trauma patients to provide information on a patient's coagulation status, particularly when the patient is requiring multiple blood products. This allows the physician to deliver a targeted hemostatic resuscitation appropriate for the patient needs in real-time. This can result in a decrease of blood products and quicker reversal of the trauma induced coagulopathy.

Riley Hospital for Children at IU Health has a TEG 5000 machine (Haemonetics Corp.) which performs the coagulation tests needed to help guide the resuscitation of a critical trauma patient. While an improvement over previous tests (such as INR, platelet count, PTT), the TEG 5000 still takes 45-60 minutes to get the results needed to guide fluid/blood resuscitation, making the results outdated as the patient has potentially received multiple units of blood products and/or had additional bleeding during that time. The TEG 5000 machine also has very specific environmental, and preparation needs (i.e. flat surface which is not bumped; controlled pipetting (dropping) of blood products into machine as well as mixing of reagents) that is very difficult to do in a busy trauma bay/emergency department with a critical patient.

The TEG 6s assays are performed in a microfluidic cartridge which only requires a small amount of a patient's blood be transferred to the cartridge for analysis. The vibration frequency of the blood meniscus at which resonance occurs is used to create a clot dynamics tracing. The sample is drawn automatically into the testing chambers rather than requiring manual pipetting, leading to less user variability. This simpler operation provides results in 15-20 minutes, making the test more clinically useful in guiding transfusion therapy during active bleeding.

TEG 6s and TEG 5000 have been evaluated in adult patients with good agreement between the modalities. More specifically, the TEG 6s has been validated in adult trauma patients. However, few pediatric studies exist.

ELIGIBILITY:
Inclusion Criteria:

-Patients less than 18 years of age undergoing elective pediatric surgical care in the operating room at Riley Hospital for Children

Exclusion Criteria:

* Known disorder of coagulation pathway(s)
* Administration of medications that may alter the coagulation cascade
* Patients in foster care or wards of the court

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
TEG 6s viscoelastic measurement, angle, in pediatric surgical patients | 2 months
  To validate the TEG 6S measurement values in pediatric patients by comparing its viscoelastic values with those existing published reference ranges
TEG 6s viscoelastic measurements, R time, in pediatric surgical patients | 2 months
  To validate the TEG 6S measurement values in pediatric patients by comparing its viscoelastic values with those existing published reference ranges
TEG 6s viscoelastic measurement, maximum amplitude, in pediatric surgical patients | 2 months
  To validate the TEG 6S measurement values in pediatric patients by comparing its viscoelastic values with those existing published reference ranges
TEG 6s viscoelastic measurement, lysis at 30 minutes, in pediatric surgical patients | 2 months
  To validate the TEG 6S measurement values in pediatric patients by comparing its viscoelastic values with those existing published reference ranges

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided